CLINICAL TRIAL: NCT00686881
Title: A Clinical Study of SCH 54031 as Monotherapy in IFN-treated Patients With Chronic Hepatitis C
Brief Title: Efficacy of Peginterferon Alfa-2b (SCH 054031) vs Glycyrrhizin in Interferon (IFN)-Treated Patients With Chronic Hepatitis C and F2/F3 Liver Fibrosis (P04773)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: This study was terminated due to low enrollment
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P04773; JPC-05-356-30
Record Dates: First submitted 2008-05-27; First posted 2008-05-30 (Estimated); Results first posted 2012-03-06 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis C, Chronic
Keywords: hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — peginterferon alfa-2b

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PegIFN-2b (Experimental): Participants receiving PegIFN-2b at 0.5 ug/kg subcutaneously (SC) once a week for up to 156 weeks.
  Interventions: Biological: Peginterferon alfa-2b (PegIFN-2b)
- SNMC (Active Comparator): Participants receiving SNMC 40 mL by intravenous (IV) injection or IV infusion 3 times weekly for up to 156 weeks.
  Interventions: Drug: Comparator: Stronger neo minophagen C (SNMC)

INTERVENTIONS:
Biological: Peginterferon alfa-2b (PegIFN-2b) — PegIFN-2b administered at a dose of 0.5 ug/kg SC once a week for 156 weeks
  Other Names: SCH 054031; Pegylated interferon alfa-2b
  Arms: PegIFN-2b
Drug: Comparator: Stronger neo minophagen C (SNMC) — SNMC (as glycyrrhizin-containing compound) administered at 40 mL by intravenous (IV) injection or IV infusion 3 times weekly for 156 weeks .
  Arms: SNMC

SUMMARY:
The objective of this study is to compare the efficacy of peginterferon alfa-2b (PegIFN-2b) monotherapy administered at a dose of 0.5 ug/kg vs stronger neo minophagen C (SNMC) in participants with chronic hepatitis C (CHC) and liver fibrosis (Metavir fibrosis score of F2 and F3) who were previously treated with interferon. The trial will evaluate the effect of treatment on the progression of liver fibrosis, liver inflammation, and liver function. Treatment will be administered for up to 156 weeks with a 4-week follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic hepatitis C previously treated with interferon
* At least 20 years of age
* Liver fibrosis score rated as F2 or F3 based on the result of liver biopsy at screening
* Female patients willing to use contraception
* Body weight from 35.0 kg to 110.0 kg (inclusive)
* Positive for hepatitis C virus ribonucleic acid (HCV-RNA) by qualitative assay
* Patients who meet the following laboratory criteria:

  * Serum alanine aminotransferase (ALT) level: >60 IU/L
  * Neutrophil count: >=1,200/mm^3
  * Platelet count: >=100,000/mm^3
  * Serum potassium level: >=3.5 mEq/L

Exclusion Criteria:

* Patients who received interferon therapy within 90 days of Screening
* Patients who have received antiviral agents or antitumor agents, or immunomodulator therapy (including chronic glucocorticoids and radiotherapy) within 90 days of Screening (excluding local administration and topical use)
* Patients who have received other investigational drugs within 90 days of Screening
* Hepatitis B surface antigen (HBs)positive
* Antinuclear antibody titer of 1:320 or higher
* Creatinine level exceeding the upper limit of the reference range measured at screening test 2;
* Fasting blood glucose level of >=126 mg/dL
* Patients on insulin therapy regardless of the fasting blood glucose level
* Patients who have a concurrent or past history of any of the following conditions: liver cirrhosis, liver failure, or liver carcinoma; hepatic encephalopathy, esophageal varices requiring treatment, or ascites; suicidal attempt or ideation; epileptic seizures requiring drug therapy; angina pectoris, heart failure, myocardial infarction or fatal arrhythmia; autoimmune disease (Hashimoto's disease [chronic thyroiditis], Crohn's disease, ulcerative colitis, rheumatoid arthritis, idiopathic thrombocytopenic purpura, systemic lupus erythematosus, autoimmune hemolytic anemia, scleroderma, etc.); malignant tumors (it is permitted to register patients with at least 5 years after cure).
* Patients who concurrently have any of the following conditions: liver disease such as autoimmune hepatitis, alcoholic liver injury, and drug-induced hepatitis; hemophilia; depression or schizophrenia which requires treatment; hypertension which cannot be controlled by drug therapy or arrhythmia which requires treatment, chronic pulmonary disease; abnormal thyroid function that cannot be controlled by drug therapy; organ transplants (other than corneal, hair transplant, etc.); aldosteronism, myopathy, or hypokalemia.
* Patients with a history of hypersensitivity to interferon preparations or biological products such as vaccines
* Patients with a history of hypersensitivity to monoammonium glycyrrhizinate, glycine, or L-cysteine monohydrochloride;
* Women who are pregnant or lactating, and women in whom pregnancy cannot be ruled out based on the result of serum human chorionic gonadotropin (HCG) measurement at Screening

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2006-12; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Groups:
- PegIFN-2b: Participants receiving peginterferon alfa-2b (PegIFN-2b) at 0.5 ug/kg subcutaneously (SC) once a week for up to 156 weeks.
- SNMC: Participants receiving stronger neo minophagen C (SNMC) 40 mL by intravenous (IV) injection or IV infusion 3 times weekly for up to 156 weeks.
Period: Overall Study
Arm/Group | PegIFN-2b | SNMC
Started | 127 (After randomization, 2 participants withdrew consent and did not receive study drug.) | 134 (After randomization, 6 participants withdrew consent and did not receive study drug.)
Completed | 45 | 53
Not Completed | 82 | 81
Not completed — Withdrawal by Subject | 11 | 18
Not completed — Lost to Follow-up | 0 | 1
Not completed — Treatment-related adverse event | 10 | 9
Not completed — Met discontinuation criteria | 5 | 0
Not completed — Onset of malignant tumor | 11 | 11
Not completed — Lack of Efficacy | 4 | 3
Not completed — Physician Decision | 1 | 0
Not completed — Circumstances of site | 1 | 1
Not completed — Did not meet protocol eligibility | 1 | 0
Not completed — Irregular visits | 1 | 0
Not completed — Study discontinuation | 35 | 32
Not completed — Never received study drug | 2 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PegIFN-2b | SNMC | Total
Number analyzed (Participants) | 125 | 127 | 252
Age, Continuous [Mean (Standard Deviation); unit: years] — Of the 261 randomized participants, 253 received study drug; 1 of these participants in the SNMC Arm had no data available after initial treatment and is excluded from study analyses.
  years | 59.8 (9.5) | 60.7 (8.9) | 60.3 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Of the 261 randomized participants, 253 received study drug; 1 of these participants in the SNMC Arm had no data available after initial treatment and is excluded from study analyses.
  Participants
    Female | 60 | 65 | 125
    Male | 65 | 62 | 127
Region of Enrollment [Number; unit: participants] — Of the 261 randomized participants, 253 received study drug; 1 of these participants in the SNMC Arm had no data available after initial treatment and is excluded from study analyses.
  participants
    Japan | 125 | 127 | 252

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Change in Metavir Fibrosis Score
Description: Metavir fibrosis score is a 5-point scale based on the amount of fibrosis in the liver, ranging from F0 (best, no fibrosis) to F4 (worst, cirrhosis).
Time Frame: Baseline and discontinuation of treatment (up to 156 weeks)
Population: All treated participants excluding 2 participants on the PegIFN-2B arm and 1 participant on the SNMC arm for whom baseline data were non-evaluable or for whom no post-baseline data were available.
Measure: Number; unit: Participants
Arm/Group | PegIFN-2b | SNMC
Number analyzed (Participants) | 123 | 126
Participants
  Participants with ≥1grade lower score (improved) | 13 | 11
  Participants with no change in score | 79 | 79
  Participants with ≥1 grade higher score (worsened) | 31 | 36

2. Secondary Outcome: Number of Participants With Alanine Aminotransferase (ALT) Normalization of >16 Weeks Duration
Description: The ALT was judged to have been normalized when the ALT level was 35 IU/L or below.
Time Frame: Week 24
Population: All treated participants except 1 SNMC participant who had no available data after initial treatment.
Measure: Number; unit: Participants
Arm/Group | PegIFN-2b | SNMC
Number analyzed (Participants) | 125 | 127
Participants | 9 | 2

3. Secondary Outcome: Number of Participants With Change in Metavir Inflammation Score
Description: Metavir inflammation score is a 4-point scale based on the severity of inflammation in the liver, ranging from A0 (best, no activity) to A3 (worst, severe activity).
Time Frame: Baseline and Week 48
Population: All treated participants excluding 3 participants on the PegIFN-2b arm and 1 participant on the SNMC arm for whom baseline data were non-evaluable or for whom no post-baseline data were available.
Measure: Number; unit: Participants
Arm/Group | PegIFN-2b | SNMC
Number analyzed (Participants) | 122 | 126
Participants
  Participants with ≥1grade lower score (improved) | 48 | 23
  Participants with no change in score | 55 | 61
  Participants with ≥1grade higher score (worsened) | 19 | 42

ADVERSE EVENTS:
Description: All treated participants except one SNMC participant who had no available data after initial treatment.
Arm/Group | PegIFN-2b | SNMC
Serious Adverse Events (participants affected / at risk) | 32/125 | 23/127
Other Adverse Events (participants affected / at risk) | 125/125 | 123/127
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PegIFN-2b (N=125) | SNMC (N=127)
IDIOPATHIC THROMBOCYTOPENIC PURPURA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
PRINZMETAL ANGINA (Cardiac disorders) | 0 (0) | 1 (1)
DEAFNESS NEUROSENSORY (Ear and labyrinth disorders) | 1 (1) | 0 (0)
MENIERE'S DISEASE (Ear and labyrinth disorders) | 1 (1) | 0 (0)
COLONIC POLYP (Gastrointestinal disorders) | 0 (0) | 1 (1)
DUODENAL ULCER (Gastrointestinal disorders) | 1 (1) | 0 (0)
GINGIVAL BLEEDING (Gastrointestinal disorders) | 1 (1) | 0 (0)
PANCREATITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
PANCREATITIS ACUTE (Gastrointestinal disorders) | 1 (1) | 0 (0)
VARICES OESOPHAGEAL (Gastrointestinal disorders) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 1 (1) | 0 (0)
APPENDICITIS (Infections and infestations) | 1 (1) | 0 (0)
BRONCHIECTASIS (Infections and infestations) | 1 (1) | 0 (0)
BRONCHOPNEUMONIA (Infections and infestations) | 1 (1) | 0 (0)
PYELONEPHRITIS (Infections and infestations) | 1 (1) | 0 (0)
PYELONEPHRITIS ACUTE (Infections and infestations) | 1 (1) | 0 (0)
SEPSIS (Infections and infestations) | 0 (0) | 1 (1)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
FRACTURED SACRUM (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
HAND FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
MENISCUS LESION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SKIN LACERATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
TENDON RUPTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
GASTRIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
HEPATIC NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8) | 10 (10)
LARGE INTESTINE CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
METASTASES TO LUNG (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OVARIAN NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
PANCREATIC CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
RECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
RENAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 1 (1) | 1 (1)
INTRAVENTRICULAR HAEMORRHAGE (Nervous system disorders) | 0 (0) | 1 (1)
LACUNAR INFARCTION (Nervous system disorders) | 1 (1) | 0 (0)
PARALYSIS (Nervous system disorders) | 0 (0) | 1 (1)
ANXIETY DISORDER (Psychiatric disorders) | 0 (0) | 1 (1)
CALCULUS URETERIC (Renal and urinary disorders) | 1 (1) | 0 (0)
PSORIASIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
ANEURYSM RUPTURED (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PegIFN-2b (N=125) | SNMC (N=127)
PALPITATIONS (Cardiac disorders) | 8 (13) | 6 (7)
ASTHENOPIA (Eye disorders) | 7 (7) | 4 (4)
CONJUNCTIVITIS (Eye disorders) | 13 (19) | 2 (2)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 16 (21) | 9 (16)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 7 (9) | 3 (4)
ABDOMINAL PAIN (Gastrointestinal disorders) | 35 (79) | 22 (32)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 14 (15) | 14 (21)
CONSTIPATION (Gastrointestinal disorders) | 32 (40) | 10 (10)
DENTAL CARIES (Gastrointestinal disorders) | 7 (10) | 8 (8)
DIARRHOEA (Gastrointestinal disorders) | 35 (63) | 17 (31)
NAUSEA (Gastrointestinal disorders) | 40 (76) | 20 (22)
PERIODONTITIS (Gastrointestinal disorders) | 8 (8) | 6 (6)
STOMATITIS (Gastrointestinal disorders) | 15 (22) | 7 (11)
TOOTHACHE (Gastrointestinal disorders) | 6 (6) | 8 (12)
VOMITING (Gastrointestinal disorders) | 9 (10) | 9 (10)
CHILLS (General disorders) | 50 (76) | 12 (14)
INJECTION SITE ERYTHEMA (General disorders) | 34 (43) | 1 (1)
INJECTION SITE PRURITUS (General disorders) | 45 (61) | 3 (4)
MALAISE (General disorders) | 97 (166) | 51 (81)
OEDEMA PERIPHERAL (General disorders) | 9 (9) | 12 (13)
PYREXIA (General disorders) | 87 (171) | 25 (36)
THIRST (General disorders) | 6 (6) | 9 (12)
CYSTITIS (Infections and infestations) | 7 (10) | 5 (7)
GASTROENTERITIS (Infections and infestations) | 4 (6) | 8 (10)
NASOPHARYNGITIS (Infections and infestations) | 77 (157) | 81 (256)
ORAL HERPES (Infections and infestations) | 7 (9) | 4 (6)
CONTUSION (Injury, poisoning and procedural complications) | 13 (18) | 6 (9)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 15 (16) | 12 (13)
TOOTH FRACTURE (Injury, poisoning and procedural complications) | 9 (10) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 34 (42) | 16 (21)
ALPHA 1 FOETOPROTEIN INCREASED (Investigations) | 4 (6) | 9 (10)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 47 (58) | 21 (26)
BASOPHIL COUNT INCREASED (Investigations) | 18 (42) | 27 (46)
BILIRUBIN CONJUGATED INCREASED (Investigations) | 5 (5) | 10 (19)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 12 (16) | 16 (24)
BLOOD BILIRUBIN INCREASED (Investigations) | 3 (3) | 8 (13)
BLOOD POTASSIUM DECREASED (Investigations) | 12 (15) | 17 (27)
BLOOD POTASSIUM INCREASED (Investigations) | 5 (6) | 8 (10)
BLOOD PRESSURE INCREASED (Investigations) | 12 (15) | 22 (28)
BLOOD THYROID STIMULATING HORMONE INCREASED (Investigations) | 29 (38) | 14 (19)
C-REACTIVE PROTEIN INCREASED (Investigations) | 16 (18) | 14 (19)
EOSINOPHIL COUNT INCREASED (Investigations) | 32 (52) | 32 (53)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 30 (37) | 23 (32)
HAEMATOCRIT DECREASED (Investigations) | 40 (60) | 10 (11)
HAEMOGLOBIN DECREASED (Investigations) | 41 (52) | 11 (13)
HYALURONIC ACID INCREASED (Investigations) | 62 (90) | 46 (70)
LYMPHOCYTE COUNT DECREASED (Investigations) | 80 (134) | 45 (107)
LYMPHOCYTE COUNT INCREASED (Investigations) | 28 (51) | 34 (69)
MONOCYTE COUNT INCREASED (Investigations) | 13 (14) | 8 (13)
NEUTROPHIL COUNT DECREASED (Investigations) | 62 (111) | 9 (12)
NEUTROPHIL COUNT INCREASED (Investigations) | 31 (48) | 50 (77)
PLATELET COUNT DECREASED (Investigations) | 74 (109) | 19 (24)
RED BLOOD CELL COUNT DECREASED (Investigations) | 41 (57) | 7 (7)
TRI-IODOTHYRONINE FREE DECREASED (Investigations) | 11 (12) | 6 (6)
WEIGHT DECREASED (Investigations) | 14 (14) | 5 (5)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 68 (104) | 9 (15)
WHITE BLOOD CELL COUNT INCREASED (Investigations) | 8 (13) | 21 (21)
DECREASED APPETITE (Metabolism and nutrition disorders) | 57 (91) | 22 (30)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 72 (123) | 31 (41)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 26 (35) | 31 (50)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 9 (16) | 13 (22)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 7 (7) | 9 (13)
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 14 (16) | 7 (7)
MYALGIA (Musculoskeletal and connective tissue disorders) | 68 (108) | 24 (39)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 10 (10) | 9 (11)
TENOSYNOVITIS (Musculoskeletal and connective tissue disorders) | 2 (2) | 8 (8)
DIZZINESS (Nervous system disorders) | 19 (25) | 15 (21)
HEADACHE (Nervous system disorders) | 82 (164) | 42 (73)
HYPOAESTHESIA (Nervous system disorders) | 8 (8) | 8 (10)
INSOMNIA (Psychiatric disorders) | 49 (78) | 15 (17)
COUGH (Respiratory, thoracic and mediastinal disorders) | 13 (19) | 15 (17)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 11 (35) | 10 (17)
OROPHARYNGEAL DISCOMFORT (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 2 (2)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 14 (28) | 12 (21)
UPPER RESPIRATORY TRACT INFLAMMATION (Respiratory, thoracic and mediastinal disorders) | 9 (12) | 11 (17)
ALOPECIA (Skin and subcutaneous tissue disorders) | 42 (51) | 3 (5)
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 9 (11) | 8 (9)
ECZEMA (Skin and subcutaneous tissue disorders) | 11 (14) | 12 (20)
PRURITUS (Skin and subcutaneous tissue disorders) | 48 (94) | 24 (33)
PRURITUS GENERALISED (Skin and subcutaneous tissue disorders) | 12 (19) | 7 (8)
RASH (Skin and subcutaneous tissue disorders) | 42 (53) | 18 (25)
HYPERTENSION (Vascular disorders) | 13 (13) | 21 (23)

LIMITATIONS AND CAVEATS:
This study was prematurely discontinued because of low enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No